CLINICAL TRIAL: NCT05522959
Title: A Single Arm Intervention Study to Assess the Role of Structured Cardio-Oncology Rehabilitation Exercise to Improve Cardiovascular Health in Early Stage Breast Cancer Survivors (CORE Study)
Brief Title: Cardio-Oncology Rehabilitation Exercise
Acronym: CORE
Status: Recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Other Study IDs: 19-5080
Record Dates: First submitted 2022-07-15; First posted 2022-08-31 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Cardiac Rehabilitation; Cardio-oncology; Cardiometabolic Health; Cardiovascular Disease Risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Women with breast cancer who are referred to the cardiac rehabilitation program at the Toronto Rehabilitation Institute will be invited to enrol in this observational study. Participants will take part in an established 16-week multimodal cardiac rehabilitation program (HEALTh program) at Toronto Rehabilitation Institute and outcome measures will be assessed before and after program participation to determine the effectiveness of the program in improving cardio metabolic health. Change in VO₂peak will be assessed using Cardiopulmonary Exercise Test (CPET). Traditional cardiac risk factors, lifestyle behaviours, exercise adherence, health-related quality of life, and fatigue will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* History of early-stage breast cancer (I-III)
* Currently receiving or have completed adjuvant therapy (i.e. chemotherapy, surgery, radiation, targeted therapies)
* Able to communicate in English

Exclusion Criteria:

* Pregnancy
* Metastatic disease (Stage IV)
* Unable or unwilling to complete cardiopulmonary exercise test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female early-stage breast cancer survivors.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary Fitness | post-intervention (16 weeks)
  VO2peak assessed using cardiopulmonary exercise test

SECONDARY OUTCOMES:
Visceral adipose tissue | post-intervention (16 weeks)
  Measured only in a subset (n=30) of participants via 1.5T MRI.
Left ventricular ejection fraction | post-intervention (16 weeks)
  Measured only in a subset (n=30) of participants via 1.5T MRI.
Native myocardial T1 time | post-intervention (16 weeks)
  Measured only in a subset (n=30) of participants via 1.5T MRI.
Left ventricular mass | post-intervention (16 weeks)
  Measured only in a subset (n=30) of participants via 1.5T MRI.
lipid profile | post-intervention (16 weeks)
  Assessed via fasting blood draw
Fasting glucose | post-intervention (16 weeks)
  Assessed via fasting blood draw
hemoglobin A1c | post-intervention (16 weeks)
  Assessed via fasting blood draw
Cancer-specific, health-related quality of life | post-intervention (16 weeks)
  Functional Assessment of Cancer Therapy (FACT) questionnaire. Minimum score = 0, maximum score = 108, with higher score representing better quality of life.
Depressive symptoms | post-intervention (16 weeks)
  Patient Health Questionnaire 9 scale. Minimum value = 0, maximum value = 27, where higher score represents more depressive symptoms.
Psychosocial Stress | post-intervention (16 weeks)
  Perceived Stress Scale (PSS). Minimum value = 0, maximum value = 56, where higher score represents more perceived stress.
Cancer-related fatigue | post-intervention (16 weeks)
  Fatigue sub-scale of the Functional Assessment of Cancer Therapy (FACT) questionnaire. Minimum score = 0, maximum score = 52, with higher score representing less fatigue.

OTHER OUTCOMES:
Smoking Status | post-intervention (16 weeks)
  Smoking assessment history questionnaire
Moderate-Intensity Physical Activity Time | averaged over 7 days post-intervention
  PiezoRx® will be worn by participants for 7 days with data used to assess moderate activity time (>100 steps per minute)
Vigorous-intensity Physical Activity | averaged over 7 days post-intervention
  PiezoRx® will be worn by participants for 7 days with data used to assess vigorous activity time (>120 steps per minute)
Physical Activity Bouts per Day | averaged over 7 days post-intervention
  PiezoRx® will be worn by participants for 7 days with data used to assess bouts of physical activity per day (greater than 10 minutes of moderate/vigorous activity)
Total daily steps | averaged over 7 days post-intervention
  PiezoRx® will be worn by participants for 7 days with data used to assess total daily steps
Self-Reported Physical Activity | post-intervention (16 weeks)
  Godin Leisure Time Physical Activity Questionnaire
Diet quality | post-intervention (16 weeks)
  Rapid Eating and Activity Assessment for Participants (REAP) questionnaire. Minimum score = 13, maximum score = 39, with a higher score indicating a higher diet quality.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Kirkham, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada